CLINICAL TRIAL: NCT04764149
Title: Efficacy and Safety of Platinum Plus Continuous Intravenous Infused 5-Fluorouracil With Low Dose and Long Term Versus Other Platinum-Based Chemotherapy in Recurrent Nasopharyngeal Carcinoma: A Case-Cohort Study
Brief Title: Platinum Plus Low-dose Long-term Continuous Intravenous Infused 5-Fluorouracil in Recurrent Nasopharyngeal Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yun-fei Xia, Department of Radiation Oncology, Sun Yat-sen University Cancer Center, Sun Yat-sen University
Other Study IDs: 2020-FXY-429
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PFll Group: Patients were treated with PFLL regimen: 5-fluorouracil intravenous infusion at 200mg/m2/d for 30 continuous days and intravenous infusion of platinum (cisplatin 70 mg/m2 or nedaplatin 80/m2 or lobaplatin 30 mg/ m2) on day 1 and day 28, every 60 days. Local treatment, molecular-targeted or immune checkpoint therapy, and supportive treatment were allowed.
- Non-PFLL Group: Patients were treated with other platinum-based chemotherapy every 21 days including: PF regimen: 5-fluorouracil at a dose of 1,000 mg/m2 daily by continuous intravenous infusion on days 1-4 and intravenous infusion of cisplatin at a dose of 80 mg/m2 on day 1. GP regimen: gemcitabine at a dose of 1,000 mg/m2 by intravenous infusion on days 1, 8, and intravenous infusion of cisplatin at a dose of 80 mg/m2 on day 1. TP regimen: paclitaxel intravenous infusion at a dose of 175 mg/m2 or docetaxel at a dose of 75 mg/m2 on day 1 and intravenous infusion of cisplatin at a dose of 75 mg/m2 on day 1. TPF regimen: paclitaxel intravenous infusion at a dose of 175 mg/m2 or docetaxel at a dose of 75 mg/m2 on day 1; cisplatin intravenous infusion at a dose of 75 mg/m2 on day 1 and continuous intravenous infusion of 5-FU at a dose of 750 mg/m2 daily on days 1-5. Local treatment, molecular-targeted or immune checkpoint therapy, and supportive treatment were allowed.

SUMMARY:
Local control rates of nasopharyngeal carcinoma are increasing, but 15% of patients still have local recurrence within 5 years after initial treatment. Systematic treatment based on chemotherapy has become the mainstream approach for recurrent nasopharyngeal carcinoma which is intolerant to local therapy. we sought to find an efficient chemotherapy regimen with high tolerance according to the characteristics of chemotherapy drugs, that is, to explore the efficacy and safety of platinum plus 5-fluorouracil with continuous intravenous infusion at a low dose for a long term.

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma (NPC) is a malignant tumor of the nasopharyngeal epithelium with high sensitivity to ionizing radiation, but failure in local control was observed in approximately 15% of patients.

Chemotherapy is the cornerstone of the treatment of recurrent NPC. Many studies were aimed at the systemic treatment of recurrent NPC, but most of them were retrospective studies or phase II trials with small samples. Platinum-containing doublet chemotherapy is generally regarded as the standard treatment for recurrent NPC. After a multicenter phase III randomized clinical trial was published in 2016, gemcitabine plus cisplatin is recommended, however, less than 60% of patients could complete the treatment in the trail. Finding a proper regimen with promising efficacy results as well as high tolerance is still a big challenge.

Cisplatin plus 5-fluorouracil (PF) is a classical regimen widely used in recurrent NPC. The continuous infusion of 5-fluorouracil with low dose was investigated in esophagus carcinoma, rectal carcinoma and prostate carcinoma with encouraging outcome and acceptable toxicity. Whereas, data of platinum containing chemotherapy with low-dose continuous infused 5-fluorouracil in recurrent NPC was absent. In this study, we aimed to investigate the antitumor activity of platinum plus low-dose long-term continuous intravenous infused 5-fluorouracil (PFLL).

ELIGIBILITY:
Inclusion Criteria:

- patients involved in our study were patients who had histologically or cytologically confirmed NPC with diagnosed recurrent NPC during 2006-2018 and receiving treatment in our hospital.

Exclusion Criteria:

* Age <18 or >70 years old

  * Pathologic type unknown or except type I-III of World Health Organization classification
  * Never underwent platinum-based chemotherapy
  * Lack of information about T classification and N classification when metastasis
  * Lost follow-up within one month from the start of treatment for metastasis
  * With other malignances

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients involved in our study were patients who had histologically or cytologically confirmed NPC with diagnosed recurrent NPC during 2006-2018 and receiving treatment in our hospital.
Sampling Method: Non-Probability Sample
Enrollment: 801 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
5-year overall survival | 5 years after diagnosis of recurrent
  The period until death is detected.

CONTACTS AND LOCATIONS:
Overall Officials: Yun-fei Xia, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Department of Radiation Oncology, Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided